CLINICAL TRIAL: NCT01202617
Title: Seroquel XR in the Long Term Treatment of Schizophrenia Focus on Affective Symptoms
Brief Title: Seroquel XR in the Long Term Treatment of Schizophrenia
Acronym: SereNIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NHU-SER-2010/1
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Relapse in Schizophrenia
Keywords: Seroquel XR; schizophrenia; relapse prevention
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenic outpatients between 18 & 70 years of age

SUMMARY:
The purpose of the study is to determine whether the Seroquel XR treatment for 6 months improves the relapse prevention in schizophrenic outpatients

ELIGIBILITY:
Inclusion Criteria:

* schizophrenic outpatients on at least 600 mg Seroquel XR treatment for at least 1 month

Exclusion Criteria:

* Severe cerebro- and cardiovascular disease, severe hepatic impairment, gravidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatients
Sampling Method: Non-Probability Sample
Enrollment: 1606 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rate of patients remained relapse free after 6 months of treatment | on the 60th day of treatment
Rate of patients remained relapse free after 6 months of treatment | on the 180th day of treatment

SECONDARY OUTCOMES:
connection between relapse and affective symptoms | on the 60th day of treatment
connection between relapse and affective symptoms | 180th day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Attila Nemeth, Principal Investigator — National Psychiatric Centre; Lilla Szabo, Study Chair — AstraZeneca; Alexandra Henringh, Study Director — AstraZeneca
Locations (61):
- Hungary (61):
  - Research Site, Baja
  - Research Site, Balassagyarmat
  - Research Site, Barcs
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Dombóvár
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Research Site, Emőd
  - Research Site, Esztergom
  - Research Site, Érd
  - Research Site, Gödöllő
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Hajdusamson-Martinka
  - Research Site, Hajdúszoboszló
  - Research Site, Heves
  - Research Site, Jánoshalma
  - Research Site, Jászberény
  - Research Site, Kalocsa
  - Research Site, Karcag
  - Research Site, Kecskemét
  - Research Site, Kétegyháza
  - Research Site, Kiskunhalas
  - Research Site, Kiskunmajsa
  - Research Site, Kistarcsa
  - Research Site, Kistokaj
  - Research Site, Komárom
  - Research Site, Kozármisleny
  - Research Site, Miskolc
  - Research Site, Nagyatád
  - Research Site, Nagykanizsa
  - Research Site, Nagykálló
  - Research Site, Nagykőrös
  - Research Site, Ny�regyhaza
  - Research Site, Pécs
  - Research Site, Pomáz
  - Research Site, Salgótarján
  - Research Site, Sátoraljaújhely
  - Research Site, Soltvadkert
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szeghalom
  - Research Site, Szekszárd
  - Research Site, Szentendre
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szigetszentmiklós
  - Research Site, Szigetvár
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Tata
  - Research Site, Tatabánya
  - Research Site, Tószeg
  - Research Site, Vác
  - Research Site, Veszprém
  - Research Site, Zalegerszeg